CLINICAL TRIAL: NCT05728541
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile and Preliminary Efficacy of SYH2043 in Patients With Advanced Malignant Tumors
Brief Title: Dose Escalation and Expansion Study of SYH2043 in Patients With Advanced Malignant Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYH2043-001
Record Dates: First submitted 2023-01-27; First posted 2023-02-15 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SYH2043 (Experimental): Patients will receive SYH2043 once everyday on day 1-21 of each 28-day cycle
  Interventions: Drug: SYH2043

INTERVENTIONS:
Drug: SYH2043 — Patients will receive SYH2043 once everyday on day 1-21 of each 28-day cycle

SUMMARY:
The aim of this study is designed to evaluate the safety, tolerability, pharmacokinetics, and preliminary antitumor activity of SYH2043 in patients with advanced malignant tumors.

DETAILED DESCRIPTION:
This study is an open-label, single-arm, multi-center Phase I clinical study, which includes four stages:

A: Dose-escalation Stage: The dose escalation stage is divided into 5 dose levels, and a Bayesian Optimal Interval Design (BOIN) including accelerated titration will be used for dose escalation.

B: PK Expansion Stage: Two or three dose groups will be selected for PK expansion; After PK extension the cohort extension study will be conducted as required, and will include 4 cohorts according to the tumor types.

C: Combination dose Escalation: This study will use a 3+3 design with up to 2 dose escalation cohorts at increasing levels.

D: According to the results of stage C, 1-2 combination doses will be selected for combination dose expansion, and Simon 2 stage was adopted for the expansion stage.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged 18-75 years (inclusive);
* 2. Histological or cytological confirmation of advanced malignant tumors;
* 3. Patients who failed or were intolerant to standard treatment or had no standard treatment, and meet the criteria as below of the corresponding stages:

  * Part A and PK Expansion Stage of part B: advanced malignant tumors;
  * Cohort extension of part B: solid tumors such as locally advanced/metastatic breast cancer, relapsed/refractory ovarian cancer, locally advanced/metastatic liver cancer, etc;
  * Part C and D: locally advanced/metastatic breast cancer with histological confirmation of ER+, HER2-;
* 4. With at least one measurable lesion according to RECIST v1.1;
* 5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1;
* 6. Life expectancy greater than 3 months;
* 7. Main organs meet the following criteria within 7 days before treatment:

  * Hematology: no component blood transfusion, human granulocyte colony-stimulating factor (G-CSF), and erythropoietin (EPO) within 2 weeks prior to the investigational drug administration
  * Absolute neutrophil count (ANC) ≥1.5×10^9/L;
  * Platelet count (PLT) ≥90×10^9/L;
  * Hemoglobin (HGB) ≥90 g/L or ≥5.6 mmol/L;
  * Renal Function: Serum creatinine ≤ 1.5×ULN or creatinine clearance rate ≥ 50 mL/min;
  * Liver function: Total bilirubin (TBIL) ≤ 1.5×ULN, or ≤ 3×ULN for patients with Gilbert syndrome; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤ 2.5×ULN, or ≤ 5×ULN in case of liver metastases;
  * Coagulation Function: Activated partial thromboplastin time (APTT)≤ 2×ULN; International normalized ratio (INR)≤ 2×ULN;
* 8. The serum pregnancy test for women of childbearing potential (WOCBP) is negative within 7 days prior to the first dose of the investigational drug. Patient and his/her spouse must agree to take adequate contraception from signing of ICF to 6 months after the last dose, during which women should be non-lactating and men should refrain from donating sperms;
* 9. Patients voluntarily participate in this clinical study, understand the study procedures and sign the ICF.

Exclusion Criteria:

* 1. Have received anti-tumor treatments such as chemotherapy, radiotherapy, endocrine therapy, targeted therapy, immunotherapy, etc. within 4 weeks before the first dose of the investigational drug;
* 2. Have received other unmarketed clinical investigational drugs or treatments within 4 weeks before the first dose of the investigational drug;
* 3. Have received major surgery (excluding needle biopsy), or severe unhealed wounds, trauma, etc. within 4 weeks before the first dose of the investigational drug in the study;
* 4. Have received glucocorticoids for systemic therapy over 7 days (Prednisone>10 mg/day or equivalent doses) or other immunosuppressant within 2 weeks before the first dose of investigational drug, and patients who need long-term use these therapies;
* 5. Have received potent inhibitors or inducers of CYP3A4 and inhibitors of P-gp within 1 weeks before the first dose of the investigational drug;
* 6. The adverse events due to previous anti-tumor treatments without recovering to Grade 1 (except for alopecia; some toxicities may be excluded as judged by the investigator) according to NCI-CTCAE v5.0;
* 7. Breast cancer patients with visceral crisis or symptomatic visceral metastasis;
* 8. With active central nervous system (CNS) metastasis and/or cancerous meningitis;
* 9. Active HBV or HCV infection (HbsAg positive and/or HBcAb positive with HBV DNA ≥ 2000 IU/mL, and HCVAb positive with HCV RNA positive), or HIV positive;
* 10. Participants with a history of severe cardiovascular disease;
* 11. Inability to swallow medications orally, or conditions that, in the judgment of the investigator, significantly affect gastrointestinal absorption;
* 12. Patients who have received a live attenuated vaccine within 2 weeks before the first use of the investigational drug or plan to receive during the study;
* 13. Other situations that the investigator considers not suitable for participating in the clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
AE | Up to approximately 3 years
  Occurrence and frequency of Adverse Event
SAE | Up to approximately 3 years
  Serious Adverse Event
DLT | At the end of Cycle 1 (each cycle is 28 days)
  Dose-limiting Toxicity (DLT)
MTD | At the end of Cycle 1 (each cycle is 28 days)
  The maximum tolerated dose (MTD) (if available)
RP2D | At the end of Stage A (approximately 1 year)
  Recommended phase 2 dose (RP2D) in stage A

SECONDARY OUTCOMES:
AUC | Up to approximately 3 years
  Area under the plasma concentration versus time curve (AUC)
Cmax | Up to approximately 3 years
  Peak Plasma Concentration (Cmax)
t1/2 | Up to approximately 3 years
  Half-life (t1/2)
Tmax | Up to approximately 3 years
  Time to peak drug concentration (Tmax)
Vz/F | Up to approximately 3 years
  Apparent volume of distribution
CL/F | Up to approximately 3 years
  Apparent clearance
pRb | Up to approximately 3 years
  Explore the relationship between phosphor-retinoblastoma protein (pRb) and efficacy
ORR | Up to approximately 3 years
  Objective Response Rate
PFS | Up to approximately 3 years
  Progression-free Survival
OS | Up to approximately 3 years
  Overall Survival
DoR | Up to approximately 3 years
  Duration of Response (DoR)
DCR | Up to approximately 3 years
  Disease Control Rate (DCR)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China